CLINICAL TRIAL: NCT01884558
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of Metformin
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0051
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Metformin; Healthy Subjects
Keywords: Isavuconazole; Pharmacokinetics; Healthy Subjects; BAL8557; BAL4815; metformin
MeSH Terms: interventions — isavuconazole; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isavuconazole and metformin (Experimental): Metformin single dose on days 1 and 8. Isavuconazole three times a day (TID) on Days 4 and 5 followed by isavuconazole once daily (QD) on Days 6-9.
  Interventions: Drug: isavuconazole; Drug: metformin

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557; BAL4815
Drug: metformin — oral
  Other Names: Glucophage®

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of a single dose of metformin. Safety and tolerability of isavuconazole will be assessed alone and in combination with metformin.

DETAILED DESCRIPTION:
Subjects will check-in to the clinic on Day -1 and remain confined through completion of the study procedures on Day 10.

A follow-up telephone call will be made on Day 16 to check on health status.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and a body mass index of 18 to 32 kg/m2, inclusive.
* QTcF must be 360 to 430 msec for males and 370 to 450 msec for females
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and serum creatinine must not be above the normal range.
* Female subject is of non-childbearing potential or if of childbearing potential must use highly effective birth control from Screening through 28 days after the end of the study. Females must not be breastfeeding or donate ova from Screening through 20 days after the end of the study.
* Male subject must be using highly effective contraception from Screening through 90 days after final study drug administration. Male subject must not donate sperm starting at Screening through 90 days after final study drug administration.

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of either Short or Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes).
* The subject has a positive result for hepatitis B surface antigen, hepatitis C antibodies at Screening or is known to be positive for human immunodeficiency virus.
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions.
* The subject is a smoker (any use of tobacco or nicotine containing products) in the last 6 months.
* The subject has had treatment with any prescribed or non-prescribed drugs in the 2 weeks prior to Day 1, with the exception of occasional use of acetaminophen up to 2 g/day.
* The subject has participated in any interventional clinical study or has received any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to Screening.
* The subject has participated in a prior study with isavuconazole.
* The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening or the subject tests positive at screening or Day -1 for alcohol or drugs of abuse.
* The subject is an employee of the Astellas Group or vendors involved in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of metformin in plasma: Area Under the Concentration-Time Curve (AUC) from the time of dosing to the last quantifiable concentration (AUClast) | Days 1 and 8 (16 plasma samples obtained from time zero to 48 hours post dose)
PK of metformin in plasma: AUC from the time of dosing to infinity (AUCinf) | Days 1 and 8 (16 plasma samples obtained from time zero to 48 hours post dose)
PK of metformin in plasma: Maximum Concentration (Cmax) | Days 1 and 8 (16 plasma samples obtained from time zero to 48 hours post dose)

SECONDARY OUTCOMES:
PK variable for isavuconazole in plasma: Trough Concentration (Ctrough) | Days 6, 9 and 10 (1 sample prior to isavuconazole dosing)
Composite of PK variables for isavuconazole in plasma: AUCtau, Cmax and tmax | Days 7 and 8 (13 samples collected per day)
  AUC during the time interval between consecutive dosing (AUCtau); the time after dosing when Cmax occurs (tmax)
Composite of PK variables for metformin in plasma: t1/2, tmax, CL/F and Vz/F | Days 1 and 8 (16 plasma samples obtained from time zero to 48 hours post dose)
  Apparent Terminal Elimination Half-life (t1/2); Apparent Body Clearance After Oral Dosing (CL/F); Apparent Volume of Distribution (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States